CLINICAL TRIAL: NCT05530057
Title: Randomized, Open Label, Multi-Center, Phase II Trial of Eribulin With or Without SB3 (Trastuzumab-biosimilar) in Patients With HER2-overexpressed Recurrent or Stage IV Breast Cancer Who Have Received at Least 2 Prior HER2-directed Regimens
Brief Title: Eribulin With or Without Trastuzumab-biosimilar in Patients With HER2-overexpressed Recurrent or Stage IV Breast Cancer
Acronym: ESPERO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1905-141-1035
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-12

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — eribulin

STUDY DESIGN:
Intervention Model Description: Arm A (Eribulin + SB3) Arm B (Eribulin monotherapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eribulin + SB3 (Experimental): - Patients will receive eribulin mesylate 1.4 mg/m2 administered I.V. with infusion over 2 to 5 minutes on days 1 and 8 of each 21-day cycle and SB3 8 mg/kg I.V. over 90 minutes on day 1 of cycle 1 . Thereafter, SB3 6 mg/kg will be infused over 30 minutes on day 1 of each subsequent 21-day cycle until progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate + Samfenet (Trastruzumab-biosimilar)
- Eribulin monotherapy (Active Comparator): - Patients will receive eribulin mesylate 1.4 mg/m2 administered I.V. with infusion over 2 to 5 minutes on days 1 and 8 of each 21-day cycle until progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate + Samfenet (Trastruzumab-biosimilar) — * Patients will receive eribulin mesylate 1.4 mg/m2 administered I.V. with infusion over 2 to 5 minutes on days 1 and 8 of each 21-day cycle and SB3 8 mg/kg I.V. over 90 minutes on day 1 of cycle 1 . Thereafter, SB3 6 mg/kg will be infused over 30 minutes on day 1 of each subsequent 21-day cycle until progression or unacceptable toxicity.
  * Dose reductions for eribulin, but not for SB3, is permitted.
  * Two dose reductions (1.1, 0.7 mg/m2) are allowed for eribulin before consideration of study treatment discontinuation. Eribulin could be continued as monotherapy if trastuzumab-similar was discontinued, and vice-versa.
  Arms: Eribulin + SB3
Drug: Eribulin Mesylate — * Patients will receive eribulin mesylate 1.4 mg/m2 administered I.V. with infusion over 2 to 5 minutes on days 1 and 8 of each 21-day cycle until progression or unacceptable toxicity.
  * Two dose reductions (1.1, 0.7 mg/m2) are allowed before consideration of study treatment discontinuation.
  Arms: Eribulin monotherapy

SUMMARY:
Optimal salvage treatment for HER2-positive breast cancer after trastuzumab and T-DM1 failure still remains to be established. We would like to investigate the efficacy and safety of combination chemotherapy of eribulin and trastuzumab as salvage treatment for HER2-Positive breast cancer after exposure to trastuzumab and T-DM1

DETAILED DESCRIPTION:
HER2-targeted therapy is the mainstay therapeutic option for the treatment of HER2 positive breast cancer patients. Even after progression on HER2-targeted therapy, HER2 remains an effective therapeutic target. In a phase III randomized clinical trial, Lapatinib plus capecitabine showed superior outcome compared to capecitabine alone in HER2 positive breast cancer patients who has progressed after trastuzumab-based therapy Moreover, ado-trastuzumab emtansine (T-DM1) showed improved progression free survival (PFS) and overall survival (OS) in HER2-positive advanced breast cancer patients previously treated with trastuzumab and a taxane.

Not only switching to a different HER2-targeted agent, but rechallenge of trastuzumab has also shown efficacy in trastuzumab failed HER2-positive breast cancer patients. In HER2-positive breast cancer patients who failed trastuzumab and lapatinib, rechallenge of trastuzumab in combination with conventional chemotherapy showed response rate of 31%, PFS of 4.9 months, and OS of 19.4 months.

Eribulin mesylate is a non-taxane inhibitor of microtubule which shows efficacy in HER2-positive breast cancer. The efficacy of eribulin and trastuzumab combination chemotherapy as first line palliative chemotherapy in HER2-positive breast cancer was identified in a phase II trial. Eribulin plus trastuzumab was an effective regimen which showed response rate of 71.2% and PFS of 11.6 months.

Currently, the first line regimen for HER2-positive metastatic breast cancer is combination therapy of pertuzumab, trastuzumab, and docetaxel as a result of the CELOPARTRA trial . After failure on pertuzumab and trastuzumab based combination chemotherapy, T-DM1 is frequently used as a 2nd line therapy. Optimal salvage treatment for HER2-positive breast cancer after trastuzumab and T-DM1 failure still remains to be established. We would like to investigate the efficacy and safety of combination chemotherapy of eribulin and trastuzumab as salvage treatment for HER2-Positive breast cancer after exposure to trastuzumab and T-DM1.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old.
* Pathologically documented breast cancer that:

  * is unresectable or metastatic
  * has confirmed HER2 positive expression (immunohistochemistry or FISH) as determined according to American Society of Clinical Oncology - College of American Pathologists guidelines evaluated at a central laboratory
  * was previously treated with trastuzumab, T-DM1 or T-Dxd, and taxane (whether in recurrent/metastatic setting or neoadjuvant/adjuvant setting).
  * Less than 4 prior lines of chemotherapy or HER2 targeted therapies for treatment in metastatic disease (<4 treatment regimens for recurrent/metastatic disease excluding adjuvant treatments)
* Documented radiologic progression (during or after most recent treatment or within 6 months after completing adjuvant therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
* Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 4.5 months after the last dose of study treatment.
* Adequate hematopoietic, renal and hepatic functions.
* Adequate hematopoietic function: Absolute granulocyte count ≥1,500/mm3, platelet≥100,000/mm3, hemoglobin≥10g/mm3
* Adequate hepatic function: total bilirubin ≤2.0mg/dL, AST/ALT ≤2 x UNL, alkaline phosphatase ≤2.5 x UNL, in case with bone metastases alkaline phosphatase ≤5 x UNL
* Adequate renal function: Serum creatinine ≤1.5mg/dL
* a left ventricular ejection fraction of 50% or more (determined by echocardiography or multiple-gated acquisition [MUGA(Multigated Blood Pool Scan)] scanning)
* CNS(central nervous system) metastasis is permitted if asymptomatic or controlled with minimal steroid requirement and is documented to be non-progressing at study entry.
* Negative result for urine or serum pregnancy tests within the screening period in premenopausal patients
* Ability to understand and comply with protocol during study period
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Prior treatment with eribulin
* Uncontrolled or significant cardiovascular disease
* History of documented congestive heart failure (CHF) or systolic dysfunction (LVEF <50%)
* High-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade Atrioventricular-block, supraventricular arrhythmias, prolonged QTc(corrected QT interval) which are not adequately rate-controlled)
* Angina pectoris requiring antianginal medication
* Clinically significant valvular heart disease
* Evidence of transmural infarction on ECG
* Poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic >100mm Hg)
* Pregnant or lactating women or women of childbearing potential, including women whose last menstrual period was ,12 months ago (unless surgically sterile) who are unable or unwilling to use adequate contraceptive measures during the study treatment period.
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer and thyroid cancer. For other types of cancer, patients could be included if there is no evidence of disease for more than 2 years.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled GI disease (e.g., Crohn's disease, ulcerative colitis)
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Concurrent disease or serious medical disorder, for example, active or uncontrolled infection, interstitial lung disease (ILD) or any psychiatric condition prohibiting understanding or rendering of informed consent.
* Patients who have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study agents or their excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint(PFS) | First day of study treatment to the date of disease progression or death due to any cause, whichever came first, assessed up to 2 years
  PFS is defined as the time from randomization to first documented disease progression as determined by the investigator using RECIST 1.1 or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Enrollment to end of treatment up to 2 years
  Objective response, defined as a CR or PR, will be determined by investigator tumor assessment using RECIST 1.1. Patients without a post-baseline tumor assessment will be considered non-responders.
Duration of objective response (DOR) | Enrollment to end of treatment up to 2 years
  DOR is defined as the time from first occurrence of a documented objective response (PR or CR) to disease progression, as determined by investigator tumor assessment using RECIST 1.1, or death from any cause, whichever occurs first
Clinical benefit rate (CBR) | Enrollment to end of treatment up to 2 years
  Clinical benefit rate, defined as having received CR or PR of any duration or stable disease (SD) ≥ 4 months per RECIST v1.1. Patients without a post-baseline tumor assessment will be considered non-responders
Overall survival (OS) | First day of study treatment to the date of death due to any cause, assessed up to 2 years
  OS is defined as the time from randomization to death from any cause. Patients who are alive as of the data cut-off date of the analysis will be censored at the last known date they were alive
Safety profile (Treatment-related adverse events as assessed by CTCAE v4.0) | First day of study treatment to end of treatment, assessed up to 2 years
  Number of participants with treatment-related adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD,PhD, Principal Investigator — Study Principal Investigato
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No